CLINICAL TRIAL: NCT06563778
Title: A Randomized, Open-label, Phase 2 Trial of Chidamide+Decitabine Plus Anti-PD-1 Antibody for Patients With R/R cHL Who Are Transplant-ineligible or Refused Transplant
Brief Title: Chidamide+Decitabine Plus Anti-PD-1 Antibody for Patients With R/R cHL Who Are Transplant-ineligible or Refused Transplant.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-089
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Ineligible Or Refused Transplant Patients With Classical Hodgkin Lymphoma
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide+Decitabine+ Anti-PD-1 Antibody (Experimental): Chidamide is a novel and orally active benzamide class of HDAC inhibitor that selectively inhibits activity of HDAC1, 2, 3 and 10, which can Induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance. Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1(DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function. Immune checkpoint inhibitors have emerged as effective therapies for many cancers by promoting the reactivation and restoring function of T cells.
  Interventions: Drug: Chidamide; Decitabine; Anti-PD-1 Antibody
- Brentuximab Vedotin+ Bendamustine+anti-PD-1 antibody (Active Comparator)
  Interventions: Drug: Brentuximab Vedotin+ Bendamustine+Anti-PD-1 antibody

INTERVENTIONS:
Drug: Chidamide; Decitabine; Anti-PD-1 Antibody — Chidamide 10mg/day, day1-4; 20mg/day, day 8,11, 15, 18. Decitabine 10mg/day, day1-5. Physicians will decide which immune checkpoint inhibitors will be used during treatment.
  Arms: Chidamide+Decitabine+ Anti-PD-1 Antibody
Drug: Brentuximab Vedotin+ Bendamustine+Anti-PD-1 antibody — Brentuximab Vedotin 1.2-1.8mg/kg day 1, Bendamustine 70-90mg/m2 day1-2, Anti-PD-1 antibody day 2. Physicians will decide which immune checkpoint inhibitors will be used during treatment.
  Arms: Brentuximab Vedotin+ Bendamustine+anti-PD-1 antibody

SUMMARY:
The prognosis for patients with relapsed/refractory classical Hodgkin lymphoma (cHL) who refuse or are ineligible for transplant is poor. This open label, randomized, phase 2 study aims to evaluate the efficacy of Chidamide+Decitabine plus Anti-PD-1 Antibody and Brentuximab Vedotin + Bendamustine plus Anti-PD-1 Antibody in transplant-ineligible or refused transplant diagnosed R/R cHL. The primary objective of the study is to evaluate progression-free survival.

DETAILED DESCRIPTION:
The prognosis of refractory or early-relapsed lymphoma is poor, and it is even worse for those who are not eligible or refuse transplantation. Although many salvage regimens have been developed, there is no standard of care. Preliminary clinical observations have shown that Chidamide +Decitabine plus Anti-PD-1 Antibody might be beneficial for these patients. Brentuximab Vedotin or Bendamustine plus Anti-PD-1 Antibody are both standard regimens.The combination of Brentuximab Vedotin, Bendamustine and Anti-PD-1 Antibody may be another effective regimen. This open-label, randomized, phase 2 study aims to evaluate the efficacy of Chidamide+Decitabine plus anti-PD-1 antibody and Brentuximab Vedotin + Bendamustine plus Anti-PD-1 Antibody, in patients with classical Hodgkin lymphoma who are transplant-ineligible or refused transplant .

The primary objective of the study is to evaluate the progression free survival. The key secondary end points are complete response rate, objective response rate and the safety.

ELIGIBILITY:
Inclusion Criteria: 1.18 to 75 years of age. 2.ECOG performance of less than 2. 3.Subjects must have histological confirmation classical Hodgkin lymphoma (cHL). 4. Patients must have at least two lines of antitumor therapy, those who were transplant-ineligible or refused transplant. 5.Life expectancy of at least 3 months. 6.Subjects with lymphoma must have at least one measureable lesion >1cm as defined by lymphoma response criteria. 7. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to ≤ grade 1 toxicity. 8.Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months. 9.Subjects must have adequate marrow, live, renal and heart functions.

-

Exclusion Criteria:1. Subjects have received the combination therapy of Chidamide+Decitabine and anti-PD-1 antibody or Brentuximab Vedotin + Bendamustine Plus Anti-PD-1 Antibody. 2.Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications. 3. Serious uncontrolled medical disorders or active infections, pulmonary infection especially. 4. Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month. 5. Prior organ allograft. 6. Women who are pregnant or breastfeeding. 7. Women with a positive pregnancy test on enrollment or prior to investigational product administration. 8. Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Time from the date of first administration of the study drug to disease progression or death from any cause (any earliest date).

SECONDARY OUTCOMES:
Complete response rate (CRR) | 1 year
  CRR assess by investigators per the 2014 Lugano classification rate of subjects achieved complete response in all evaluable subjects
Objective response rate (ORR) | 1 year
  The percentage of patients with CR or PR was determined according to the revised lymphoma efficacy evaluation criteria (Lugano 2014 criteria).
Number of Subjects with treatment-related adverse events (AEs) | 1 year
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0

OTHER OUTCOMES:
Biomarkers predictive of efficacy and toxicity | 1 year
  Biomarkers such as PD-1 from tumor tissue and peripheral blood will be assessed for their potential in predicting clinical efficacy and toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China